CLINICAL TRIAL: NCT06372678
Title: A Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of CM326 in Participants With Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: Study of CM326 in Participants With Chronic Rhinosinusitis With Nasal Polyposis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326-102102
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 220 mg Group (Experimental): CM326 220 mg, subcutaneous (SC)
  Interventions: Biological: CM326
- 440 mg Group (Experimental): CM326 440 mg, subcutaneous (SC)
  Interventions: Biological: CM326
- placebo (Placebo Comparator): matched placebo, subcutaneous (SC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM326 — CM326 injection
  Arms: 220 mg Group; 440 mg Group
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled Phase II study to evaluate the efficacy and safety of CM326, and to observe the Pharmacokinetics, Pharmacodynamics and immumogenicity of CM326 in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP).

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a chronic inflammatory disease of the sinus mucosa. Chronic rhinosinusitis can be clinically divided into chronic rhinosinusitis without nasal polyps (CRSsNP) and chronic sinusitis with nasal polyps (CRSwNP), with an incidence ratio between the two of about 4:1. Patients with CRSwNP usually show more severe clinical symptoms and are more likely to relapse after surgery. The overall prevalence of chronic rhinosinusitis in our country is 8%, of which 11.2% are accompanied by asthma. The prevalence of chronic rhinosinusitis with nasal polyps (CRSwNP) is 1.1%. With changes in the living environment and acceleration of urbanization in China, the overall morbidity is estimated to keep rising.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 18 and 75 years old (inclusive).
* Subjects who are capable of understanding the nature of the study and voluntarily signing the Informed consent form (ICF).
* Prior treatment with systemic corticosteroids (SCS) within two years before screening, and/or contraindicate to or intolerance to systemic corticosteroids, and/or with prior surgery to nasal polyps 6 months before the screening.

Exclusion Criteria:

* Allergic or intolerant to mometasone furoate spray or CM326.
* Have received allergen-specific immunotherapy that initiated within 3 months prior to randomization or planned to be initiated during the study period.
* Participated study of CM326.
* Systemic immunosuppressive therapy for inflammatory or autoimmune diseases within 8 weeks or 5 half-lives prior to baseline (whichever is longer).
* Starting leukotriene receptor antagonist therapy within 4 weeks prior to baseline.
* With antrochoanal polyps.
* With severe deviation of the nasal septum occludes at least one nostril.
* With persistent rhinitis medicamentosas.
* With acute sinusitis, nasal infection, or upper respiratory tract infection at screening.
* Have symptoms or whose CT scan suggests allergic fungal sinusitis.
* With malignant or benign neoplasm of nasal cavities.
* With other uncontrolled serious diseases or recurrent chronic diseases.
* Have severe hepatic and renal impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of nasal polyp score (NPS) in eosinophilic chronic rhinosinusitis with nasal polyps (CRSwNP) at week 24. | Up to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality, China